CLINICAL TRIAL: NCT01297257
Title: DELIVER Study: DELiverability of the Resolute Integrity Stent in All-Comer Vessels and Cross-OvER Stenting
Acronym: DELIVER
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: IP992
Record Dates: First submitted 2010-12-20; First posted 2011-02-16 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Stent implantation — Single arm, open label stent implantation

SUMMARY:
The primary objective of the DELIVER Study is to assess the deliverability of the Resolute Integrity Stent as primary stent or as a secondary cross-over stent following delivery failure of another stent type in real world patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum legal age (18)
* Acceptable candidate for treatment with a drug-eluting stent in accordance with applicable guidelines
* Patient has consented to participate and authorized in writing the collection and release of medical information

Exclusion Criteria:

* Pregnancy
* Participating in another study that interferes with study endpoints
* Untreatable hypersensitivity or allergies to aspirin, heparin, clopidogrel, zotarolimus or similar drugs or contrast media
* Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with symptomatic ischemic heart disease due to stenotic lesions in coronary arteries or bypass graft that are amenable to percutaneous treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7845 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis Ziekenhuis, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 163 centres in Europe, Asia, the Middle East, and Latin America from January 2011 to May 2012.
Pre-assignment Details: 7845 subjects enrolled in this study. 22 Subjects removed from database, per center request. Reasons varied per center.
  83 patients had very limited data available which resulted in the inability to be included in the analysis.
Groups:
- Group 1 Resolute Integrity™ Stent Primary Stent: A total of 7740 subjects were included in the intention-to-treat analysis. These subjects had 10,499 lesions which were treated with 12,165 stents.
Period: Overall Study
Arm/Group | Group 1 Resolute Integrity™ Stent Primary Stent
Started | 7740
Completed | 7740
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1 Resolute Integrity™ Stent Primary Stent
Number analyzed (Participants) | 7740
Age, Categorical [Number; unit: participants] — Age of 20 (0.26%) patients not reported by investigators.
  participants
    <=18 years | 0
    Between 18 and 65 years | 4058
    >=65 years | 3662
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of 20 (0.26%) patients not reported by investigators
  years | 63.5 (11.2)
Gender [Number; unit: participants] — Gender of 20 (0.26%) patients not reported by investigators
  participants
    Female | 1858
    Male | 5862

OUTCOME MEASURES:

1. Primary Outcome: Delivery Success
Description: The primary endpoint for this study is delivery success defined as complete passage of the Resolute Integrity stent across the target lesion with full expansion of the stent to the desired diameter at the desired location.
Time Frame: stent implantation until hospital discharge (average 1-3 days)
Measure: Number; unit: stents
Units Other Than Participants: Stents
Groups:
- Group 1 Resolute Integrity™ Stent Primary Stent: A total of 7,740 subjects were included in the intention-to-treat analysis. These subjects had 10,499 lesions which were treated with 10,733 Resolute Integrity™ Stents
Arm/Group | Group 1 Resolute Integrity™ Stent Primary Stent
Number analyzed (Participants) | 7740
Number analyzed (Stents) | 10733
stents | 10617

2. Secondary Outcome: In-hospital MACE (Major Adverse Cardiac Event)
Time Frame: stent implantation until hospital discharge (average 1-3 days)
Measure: Number; unit: Participants
Arm/Group | Group 1 Resolute Integrity™ Stent Primary Stent
Number analyzed (Participants) | 7740
Participants | 126

ADVERSE EVENTS:
Time Frame: stent implantation until hospital discharge (average 1-3 days)
Arm/Group | Group 1 Resolute Integrity™ Stent Primary Stent
Serious Adverse Events (participants affected / at risk) | 126/7740
Other Adverse Events (participants affected / at risk) | 0/7740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Resolute Integrity™ Stent Primary Stent (N=7740)
Death (General disorders) | 19 (19) — All Death 0.2% (19/7740) Cardiac Death 0.2% (15/7740)
Major Adverse Cardiac Event (Cardiac disorders) | 126 (126) — Defined as in-hospital death, myocardial infarction (Q-wave and non Q-wave), emergent coronary bypass surgery, or repeat target lesion revascularization (clinically driven/clinically indicated) by percutaneous or surgical method
Myocardial Infarction (Cardiac disorders) | 103 (103)
Definite/Probable Stent Thrombosis (Injury, poisoning and procedural complications) | 14 (14) — According to Academic Research Consortium (ARC) Definition for Stent Thrombosis
Clinically-driven Target Lesion Revascularization (Surgical and medical procedures) | 10 (10) — Revascularization at target lesion (TL) with positive functional ischemia study/ischemic symptoms AND angiographic minimal lumen diameter stenosis >=50%, or revascularization of TL with diameter stenosis >=70% without angina/positive functional study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For any publication or presentation of the Protected Materials or any portion thereof, a manuscript of the paper, abstract or other materials will be provided by Consultant to Sponsor for its approval at least sixty (60) days for manuscripts and thirty (30) days for presentations prior to outside submission. Medtronic shall have the right to request reasonable modifications of any manuscript or other materials to be published or presented.